CLINICAL TRIAL: NCT03013322
Title: Anticholium® Per Se a Randomized, Double-blind, Placebo-controlled, Monocentric Trial on the Adjunctive Use of Physostigmine Salicylate (Anticholium®) in Perioperative Sepsis and Septic Shock
Brief Title: Anticholium® Per Se
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Johannes Zimmermann, Dr. med. Johannes B. Zimmermann, MSc, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D.10060224
Record Dates: First submitted 2017-01-01; First posted 2017-01-06 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Shock, Septic; Sepsis; Perioperative Period
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Physostigmine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Active Comparator): The treatment group receives an infusion of 0.04 mg/kg physostigmine salicylate with a maximum dose of 4 mg. The infusion is administered at 0.4 mg/min (= 1 mL/min = 60 mL/h). The initial dose is followed by a continuous infusion of 0.017 mg/min, i.e. 1 mg/h (= 0.042 mL/min = 2.5 mL/h) for 2-5 days, i.e. 48-120 hours (treatment phase).
  Interventions: Drug: Physostigmine
- Placebo Group (Placebo Comparator): The placebo group is treated with 0.9% sodium chloride.
  Interventions: Drug: Isotonic Saline

INTERVENTIONS:
Drug: Physostigmine
  Other Names: Anticholium
  Arms: Treatment Group
Drug: Isotonic Saline
  Arms: Placebo Group

SUMMARY:
Anticholium® per Se is a randomized, double-blind, placebo-controlled, monocentric trial to assess whether the CAP can be transferred from bench to bedside. In this pilot study, 20 patients with perioperative sepsis and septic shock as a result of intra-abdominal infection are enrolled. According to randomization, participants are treated with physostigmine salicylate (verum group) or 0.9% sodium chloride (placebo group) for up to 5 days. The mean Sequential Organ Failure Assessment (SOFA) score during treatment and subsequent intensive care of up to 14 days is used as surrogate outcome (primary endpoint). Secondary outcome measures include 30- and 90-day mortality. An embedded pharmacokinetics and pharmacodynamics study investigates plasma concentrations of physostigmine and its metabolite eseroline. Further analyses will contribute to the understanding of the role of various cytokines in the pathophysiology of human sepsis. A computer-generated list is used for blocked randomization.

ELIGIBILITY:
Inclusion criteria

* Age 18-85 years
* APACHE II score <34
* Intra-abdominal infection

  * findings of diffuse peritonitis or a circumscribed abscess
* Perioperative sepsis

  * and secure evidence of infection, clinically backed up or secured microbiologically
  * ≥2 of the following four criteria:

    * fever ≥38.0° C or hypothermia ≤36.0° C secured by rectal intravesical or intravascular measurement
    * tachycardia ≥90/min
    * tachypnea ≥20/min or hyperventilation secured by arterial blood gas analysis with PaCO2 ≤4.3 kPa or 33 mmHg or mechanical artificial respiration
    * leukocytosis ≥12,000/mm³ or leukopenia ≤4000/mm³ or ≥10% immature neutrophils in the differential count
* Shock (<24 h duration): necessary use of vasopressors despite adequate fluid resuscitation to keep systolic blood pressure ≥90 mmHg or mean blood pressure ≥70 mmHg
* No more than one planned and/or one emergency basis/as an emergency procedure performed since admission (no repeated revisions)
* No infaust prognosis of a primary or concomitant illness, expecting the death within the follow-up phase
* No do-not-resuscitate order
* Written informed consent of full-age patients/their legal guardian to participate [written consent (according to AMG § 40 (1) 3b)] and unable to consent adults [§ 41 (1) 2 AMG)]

Exclusion criteria

* Known hypersensitivity to physostigmine salicylate, sodium metabisulfite, sodium EDTA, or any of the other ingredients of Anticholium®
* Known contraindications against Anticholium®: gangrene, coronary artery disease
* Known absolute contraindications against Anticholium®: myotonic dystrophy; depolarization block by depolarizing muscle relaxants; intoxication by "irreversibly acting" cholinesterase inhibitors; closed craniocerebral trauma; obstruction in the gastrointestinal tract (mechanical constipation); obstruction in the urinary tract (mechanical urinary retention)
* Known relative contraindications against Anticholium®: bronchial asthma; bradycardia; AV-conduction disturbances
* Having undergone splenectomy
* Having undergone solid organ transplantation
* Positive pregnancy test, pregnancy, and lactation
* Participation in another clinical trial, according to AMG or the follow-up phase of another study, according to AMG

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2017-02-18 (Actual); Study Completion 2017-02-18 (Actual)

PRIMARY OUTCOMES:
mean Sequential Organ Failure Assessment (SOFA) score | up to 14 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h after continuous infusion is commenced
  The mean SOFA score (at least two individual values) during treatment and subsequent intensive care of up to 14 days is used as surrogate outcome in critically ill patients with perioperative sepsis and septic shock due to intra-abdominal infection.

SECONDARY OUTCOMES:
duration of artificial ventilation | up to 90 d
duration of intensive care | up to 90 d
length of stay | up to 90 d
30-day mortality | 30 d
90-day mortality | 90 d
arterial blood gas analyses | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
central venous blood gas analyses | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
partial pressure of arterial oxygen (PaO2) | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
fraction of inspired oxygen (FiO2) | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
platelet count | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
leukocyte count | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
creatinine | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
urea | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
total bilirubin | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
C-reactive protein | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
prothrombin time | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
D-dimer | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
procalcitonin | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
IL-6 | up to 30 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 14 d±8 h, 28 d±8 h, 30 d±8 h after continuous infusion is commenced
thrombin-antithrombin complex | up to 30 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 14 d±8 h, 28 d±8 h, 30 d±8 h after continuous infusion is commenced
mean blood pressure | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
frequency of vasopressors | up to 90 days
duration of vasopressors | up to 90 days
frequency of renal replacement therapy | up to 90 days
duration of renal replacement therapy | up to 90 days
Glasgow Coma Scale (GCS) score | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
Acute Physiology And Chronic Health Evaluation (APACHE) II score | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
Simplified Acute Physiology Score (SAPS) II score | up to 90 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h, 7 d±4 h, 8 d±8 h, 9 d±8 h, 10 d±8 h, 11 d±8 h, 12 d±8 h, 13 d±8 h, 14 d±8 h, 28 d±8 h, 30 d±8 h, 84 d±8 h, 90 d±8 h after continuous infusion is commenced
occurrence of side effects | up to 6 d, assessed 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h after continuous infusion is commenced
  nausea or vomiting, clinically relevant changes in heart rate or blood pressure (mainly hypotension), and clinically relevant changes in airway resistance (mainly bronchiospasms as a result of hypersensitivity reactions to the sodium metabisulfite contained in the investigational medicinal product spontaneous breathing: acute dyspnea or artificial ventilation: clinically relevant decline in respiratory volume at constant pressure settings, or clinically relevant incline in peak or inspiratory pressures at constant respiratory volumes)

OTHER OUTCOMES:
microbiological analyses of potential pathogens including susceptibility tests | up to 90 days
plasma concentrations of physostigmine | up to 6 d, assessed 3±2 min after study med, end of initial ±2 min, 10, 20, 30±2 min, 1 h±10 min, 2 h±30 min, 24, 48, 72, 96, 120±2 h after continuous (end of study med), 10, 20, 30±2 min, 1, 2 h±10 min after end of study med, 6 d ± 4 h after continuous
  determined with a validated high-performance liquid chromatography (HPLC) method
plasma concentrations of eseroline | up to 6 d, assessed 3±2 min after study med, end of initial ±2 min, 10, 20, 30±2 min, 1 h±10 min, 2 h±30 min, 24, 48, 72, 96, 120±2 h after continuous (end of study med), 10, 20, 30±2 min, 1, 2 h±10 min after end of study med, 6 d ± 4 h after continuous
  determined with a validated high-performance liquid chromatography (HPLC) method
acetylcholinesterase activity | up to 6 d, assessed 1 h±10 min, 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h after continuous infusion is commenced
  determined with ChE check mobile (Securetec, Neubiberg, Germany) from remaining material drawn for routine blood gas analyses (arterial samples)
butyrylcholinesterase activity | up to 6 d, assessed 1 h±10 min, 2 h±30 min, 24±2 h, 48±2 h, 72±2 h, 96±2 h, 120±2 h, 6 d±4 h after continuous infusion is commenced
  determined with ChE check mobile (Securetec, Neubiberg, Germany) from remaining material drawn for routine blood gas analyses (arterial samples)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes B Zimmermann, MD, MSc, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pinder N, Zimmermann JB, Gastine S, Wurthwein G, Hempel G, Bruckner T, Hoppe-Tichy T, Weigand MA, Swoboda S. Continuous infusion of physostigmine in patients with perioperative septic shock: A pharmacokinetic/pharmacodynamic study with population pharmacokinetic modeling. Biomed Pharmacother. 2019 Oct;118:109318. doi: 10.1016/j.biopha.2019.109318. Epub 2019 Aug 6. PMID 31398669
- [Derived] Pinder N, Bruckner T, Lehmann M, Motsch J, Brenner T, Larmann J, Knebel P, Hoppe-Tichy T, Swoboda S, Weigand MA, Hofer S, Zimmermann JB. Effect of physostigmine on recovery from septic shock following intra-abdominal infection - Results from a randomized, double-blind, placebo-controlled, monocentric pilot trial (Anticholium(R) per Se). J Crit Care. 2019 Aug;52:126-135. doi: 10.1016/j.jcrc.2019.04.012. Epub 2019 Apr 9. PMID 31035187
- [Derived] Zimmermann JB, Pinder N, Bruckner T, Lehmann M, Motsch J, Brenner T, Hoppe-Tichy T, Swoboda S, Weigand MA, Hofer S. Adjunctive use of physostigmine salicylate (Anticholium(R)) in perioperative sepsis and septic shock: study protocol for a randomized, double-blind, placebo-controlled, monocentric trial (Anticholium(R) per Se). Trials. 2017 Nov 10;18(1):530. doi: 10.1186/s13063-017-2231-x. PMID 29126416